CLINICAL TRIAL: NCT05490641
Title: Personalized Feedback of Wearable Biological Sensor Data to Promote Active Living in Cancer Survivors
Brief Title: Know and Own Your Movement-related Metrics Via Wearable Devices
Acronym: Project KNOWN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: American Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Yue Liao, Assistant Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0177
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Survivorship
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biofeedback Group (Experimental)
  Interventions: Behavioral: Glucose-based biofeedback
- Standard Care Group (Active Comparator)
  Interventions: Behavioral: Standard feedback

INTERVENTIONS:
Behavioral: Glucose-based biofeedback — Participants will wear a Fitbit activity tracker and receive personalized text messages over a 12-week period. During the first 4 weeks of the study period, participants will also wear a continuous glucose monitor to check their glucose levels in real-time and receive text messages based on their activity and glucose data.
  Arms: Biofeedback Group
Behavioral: Standard feedback — Participants will wear a Fitbit activity tracker and receive non-personalized text messages over a 12-week period.
  Arms: Standard Care Group

SUMMARY:
This study aims to promote daily physical activity in cancer survivors who are at high risk for type 2 diabetes (T2D) by using a personalized biological-based feedback strategy. T2D is one of the most common co-occurring conditions in cancer survivors and can worsen cancer-related health outcomes, especially in those who are insufficiently active. The investigators hypothesize that seeing the immediate impacts of exercise on their biological status will motivate cancer survivors to exercise. The investigators will use real-time data from continuous glucose monitor to demonstrate the acute impact of physical activity and measure daily activity levels using wearable trackers. As wearable sensor technology is constantly advancing, this study is the first step to exploring how researchers can use wearable sensors to help people make a direct connection between their daily behaviors and health outcomes.

DETAILED DESCRIPTION:
Physical activity plays an important role in energy balance and obesity, which is an independent risk factor for cancer recurrence and mortality. It has been estimated that cancer survivors who increased their physical activity from pre- to post-diagnosis by any level had a 39% risk reduction in total mortality. This study will use an innovative approach to motivate cancer survivors to adopt and maintain an active lifestyle and will explore a novel mediator (daily glucose pattern) of the association between physical activity and cancer-related biomarkers. Study participants will be randomly assigned into (1) a group that receives personalized biological feedback related to physical activity behaviors; and (2) a control group that receives standard educational material. The feasibility and preliminary efficacy of this wearable sensor-based, biofeedback-enhanced 12-week physical activity intervention will be evaluated. This study will provide data regarding the preliminary efficacy of using biological feedback to increase physical activity and identifying daily glucose patterns that might link to cancer-related biomarkers.

The overall goals for this study are: (1) to test the preliminary effect of a remotely delivered physical activity intervention that incorporates personalized biological-based feedback on daily physical activity levels, and (2) to explore the association between daily glucose patterns and cancer-related insulin pathway and inflammatory biomarkers in cancer survivors who are at high risk for type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older
* have had a diagnosis of cancer
* have completed curative-intended treatment for at least 3 months (except hormone therapy or long-term maintenance chemotherapy)
* be at high-risk for type 2 diabetes based on the American Diabetes Association Type 2 Diabetes Risk Test
* currently insufficiently active
* capable of participating in moderate-vigorous intensity unsupervised exercise
* have no current diagnosis or history of type 1 or 2 diabetes
* able to speak, read, and write in English
* have a smartphone with daily internet access

Exclusion Criteria:

* currently taking oral antidiabetic agents (OADs)
* current treatment with any insulin regimen other than basal insulin, e.g. prandial or pre-mixed insulin
* currently pregnant
* on dialysis
* have self-reported health issues that limit physical activity
* work overnight shifts
* unwilling to use the study devices
* current participation in other exercise or weight loss-related program or intervention
* currently on a low-carb diet
* current use of other implanted medical devices such as pacemakers
* do not have a smartphone that is compatible with the Fitbit and the LibreLink apps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of delivering personalized glucose-based feedback | Through study completion, an average of 3 months.
  The intervention will be considered feasible if ≥ 80% of participants in the intervention group are adherent to the self-monitoring protocol and ≥ 80% of participants complete the post-intervention assessment.

SECONDARY OUTCOMES:
Changes in daily physical activity level | Through study completion, an average of 3 months.
  A blinded accelerometry device will be used to measure physical activity before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Liao, MPH, PhD, Principal Investigator — University of Texas at Arlington
Locations (1):
- The University of Texas at Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liao Y, Schembre SM, Brannon GE, Pan Z, Wang J, Ali S, Beg MS, Basen-Engquist KM. Using wearable biological sensors to provide personalized feedback to motivate behavioral changes: Study protocol for a randomized controlled physical activity intervention in cancer survivors (Project KNOWN). PLoS One. 2022 Sep 13;17(9):e0274492. doi: 10.1371/journal.pone.0274492. eCollection 2022. PMID 36099282